CLINICAL TRIAL: NCT01123447
Title: A Prospective Randomized Trial Comparing Open Reduction and Internal Fixation With Non-operative Treatment for Ulnar Shaft Fractures
Brief Title: Surgical Treatment Versus Non-surgical Treatment of Ulnar Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Orthopaedic Research Legacy (Unknown); Canadian Orthopaedic Trauma Society (Other); Calgary Surgical Research Development Fund (Other); AO Research Fund (Other)
Responsible Party: Principal Investigator, Paul Duffy, Division Head, Orthopaedic Trauma, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB14-2004
Record Dates: First submitted 2010-05-10; First posted 2010-05-14 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Fracture; Trauma; Ulna Fracture; Orthopedic; Surgery
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries; Ulna Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Active Comparator): Isolated ulnar shaft fractures will be treated with open reduction and internal fixation using a limited contact dynamic compression (LC-DC) plate with screws. These will remain at the fracture site for the lifetime of the patient.
  Interventions: Procedure: Open reduction and internal fixation
- Short arm cast (Active Comparator): Those individuals randomized to the non-operative treatment group will be treated with a closed reduction and short-arm (below-elbow) cast.
  Interventions: Procedure: Closed reduction and short-arm cast

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Patients will undergo surgery for open reduction of the fracture and internal fixation with an LC-DC plate and screw fixation.
  Other Names: Limited contact dynamic compression plate (LC-DC) with screw fixation
  Arms: Surgery
Procedure: Closed reduction and short-arm cast — Patient will undergo a closed reduction and be placed in a short-arm (below-elbow) cast for 6 weeks.
  Arms: Short arm cast

SUMMARY:
The purpose of this study is to determine if surgery using a plate and screws to fix a forearm fracture (ulnar shaft) will improve functional outcome compared to non-operative treatment out to 1 year of follow-up. It is hypothesized that in skeletally mature patients with isolated ulnar shaft fractures, the patients treated with surgery will have improved functional outcomes compared to non-surgical treatment with below-elbow cast at 1-year follow-up. This will be measured by the Disabilities of the Arm, Shoulder and Hand (DASH) scores. Secondary outcomes will include SF-36, range of motion, pain, grip strength, return to work, and time to union.

DETAILED DESCRIPTION:
Ulnar diaphyseal, or "nightstick", fractures are uncommon, but fraught with complications (Pollock et al., 1983; Grace & Witmer, 1980, Atkin et al., 1995) and may prevent return to work (Atkin et al., 1995). 3 systematic reviews have concluded that there is insufficient evidence to guide treatment of isolated ulnar shaft fractures (Handoll & Pearce, 2000; Mackay et al., 2000; Bhandari & Schemitsch, 2004) and there has been no comparison between operative and non-operative management. Therefore, there is true clinical equipoise regarding optimal treatment of these injuries.

The aim of this study is to determine if open reduction and internal fixation (ORIF) is more efficacious than closed reduction and below-elbow casting for 6 weeks in restoring function of the forearm and wrist.

We hypothesize that in skeletally mature patients with isolated ulnar shaft fractures, ORIF will improve functional outcomes compared to non-operative treatment with below-elbow cast at 1-year follow-up.

The primary objective is to compare Disabilities of the Arm, Shoulder and Hand (DASH) scores at 1-year post-injury. Secondary outcome measures include SF-36, range of motion, pain, grip strength, return to work and time to union.

The study design is a multi-centre, open-label parallel randomized clinical trial. 100 skeletally mature patients with closed, extra-articular isolated ulnar diaphyseal fractures will be randomized to one of the two treatment arms. Polytrauma patients or those with pre-existing bone pathology will be excluded. Post-treatment follow-up evaluation will occur at 2, 6 and 12 weeks and at 6 and 12 months. Interim analysis will be completed by an independent Data Safety and Monitoring Committee to ensure patient safety.

Radiologic displacement, angulation and time to union will be evaluated by two independent, blinded observers. Time to fracture union will be defined as bridging callus across the fracture line on 2 views.

The sample size was calculated as 50 patients per group. Independent samples t-test will be used to compare the DASH and SF-36 scores and return to work. An ANOVA will be used for the DASH, SF-36 and range of motion comparison at each follow-up.

There is true clinical equipoise regarding optimal treatment for isolated ulnar diaphyseal fractures, therefore, the results of this trial will provide robust evidence for clinical decision-making in the treatment of these injuries by orthopaedic surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years of age and skeletally mature
* Subject has an isolated extra-articular ulnar diaphyseal fracture
* Subject presents within 14 days or less between injury and study recruitment
* Patient must be medically fit for anesthesia
* Subject is willing and able to provide written informed consent for trial participation
* Subject is willing and able to comply with the study protocol including return for all follow-up evaluations
* Subject has an isolated ulnar diaphyseal fracture (AO type 22A1.1, 22A1.2, 23A1.2, 23A1.3, 22B1.1, 22B1.2) without extension to the articular surface
* Fracture is displaced, but displacement is <50% after closed reduction, if closed reduction is required
* Fracture less than 30-degrees of angulation following closed reduction, if closed reduction is required

Exclusion Criteria:

* Subject has a pre-existing ipsilateral wrist injury, degenerative condition, or congenital anomaly
* Subject has a delay in treatment greater than 14 days from time of injury
* Subject has an active infection in the area of surgical approach
* Subject has concomitant injury which, in the opinion of the attending surgeon, is likely to impair rehabilitation or prolong ulnar fracture healing time (another long bone fracture, ipsilateral limb injury)
* Subject has a history of rheumatoid arthritis, fibrous dysplasia, chronic renal failure, Paget's disease, or osteopetrosis
* Subject has a high risk of death from surgery (ASA physical status Class V)
* Subject is likely unable to maintain follow-up (no fixed address, plans to move out of town in the next year, states unable to comply with protocol, etc)
* Subject has cognitive impairment or language difficulties that would impeded the valid completion of questionnaires
* Subject is pregnant
* Subject is a prisoner, currently detained
* Subject has an articular fracture (AO Type 23A1.1, 23B or 23C)
* Open ulnar fracture (any Gustilo grade)
* Segmental fracture
* Fractures within 2 cm of the distal radioulnar joint (AO 23A1.1)
* Fracture of the proximal 1/3 of the ulnar shaft (i.e. Monteggia fracture pattern, AO Type 21A, 22A1.3, 22B1.3)
* Pathologic fracture

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-07-02 (Actual); Primary Completion 2023-03-08 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (The DASH) | 1 year
  30-item, self-reported questionnaire that evaluates function of the affected upper extremity and will reveal the impact of the forearm injury on the function of the entire limb

SECONDARY OUTCOMES:
Range of Motion | 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  An evaluation of the range of motion about the wrist and the elbow for both the affected limb and the unaffected limb post-treatment. It will be evaluated starting at 2 weeks for the surgical group and at 6 weeks for the below-elbow cast group.
Grip Strength | 6 weeks, 12 weeks, 6 months, 12 months
  An evaluation of the grip strength for both the affected limb and the unaffected limb post-treatment.
Radiologic outcome - time to union (fracture healing) | baseline, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  Radiologic outcome will be evaluated based on bridging callus evident on 2 x-ray views (AP and lateral). Time to union will be defined as bridging callus evide on 2 x-ray views.
SF-36 | baseline, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  36-item, self-reported questionnaire is an outcome tool that examines patient-reported overall health and ease of activities of daily living
Pain Visual Analogue Score | baseline, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  • A standardized pain visual analogue scale will be used to rate pain with various activities of daily living on a scale from 0-10
DASH score | baseline, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months
  30-item, self-reported questionnaire that evaluates function of the affected upper extremity and will reveal the impact of the forearm injury on the function of the entire limb

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Duffy, MD, Principal Investigator — University of Calgary
Locations (9):
- Canada (8):
  - Dr. Paul J Duffy, Calgary, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Memorial University, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- North Bristol NHS Trust, Bristol, United Kingdom